CLINICAL TRIAL: NCT01951794
Title: CIDRZ 1225 - Validation of a Community Survey Methodology for Measuring PMTCT Program Impact
Brief Title: Validation of a Community Survey Methodology for Measuring PMTCT Program Impact
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: CIDRZ 1225; R01HD075131-01 (NIH)
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: HIV
Keywords: HIV infected; HIV exposed; HIV-free

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — We will collect Dried Blood Specimens (DBS) from both mother and infant and link them using pre-printed bar codes. For a mother who refuses real-time testing, but agrees to collection of this maternal DBS specimen, she will be provided a card with a unique study-generated identification number that can be used pick-up results at the community's designated health facility. For those who agreed to on-site HIV testing, we will retain the DBS specimens for quality assurance purposes. As part of the informed consent process, participants will also be asked whether leftover specimens may be used for future use, pending local and international ethical approvals for specified substudies.
Oversight: Data Monitoring Committee: No

SUMMARY:
Validate a promising community survey methodology for evaluating the Prevention of Mother to Child Transmission (PMTCT) program effectiveness against a "gold standard" cohort design and to identify individual- and facility-level characteristics associated with HIV-free survival among HIV-exposed infants.

DETAILED DESCRIPTION:
The overarching aim of this study is to determine the accuracy and reliability of a household survey methodology to measure PMTCT program impact. If appropriately validated, this approach could be used to monitor program effectiveness across a wide range of settings, both as part of Demographic and Health Surveys (DHS) or in stand-alone evaluations.

Specific objectives

Objective 1: To validate the community survey methodology for measuring PMTCT program effectiveness. Across 42 communities in rural Lusaka Province, we will estimate HIV-free survival among HIV-exposed children using two methodologies at the community level: a survey approach and a "gold standard" cohort approach.

Hypothesis: HIV-free survival measurements from the two study components will demonstrate strong correlation and high inter-method agreement, thus confirming the validity of the community survey for PMTCT evaluation.

Objective 2: To identify individual- and facility-level characteristics associated with HIV-free survival among HIV-exposed infants. We will determine key characteristics associated with optimal PMTCT program effectiveness, thus providing an objective measurement of "best practices" in our setting.

Hypothesis: High PMTCT service utilization and high antenatal care quality will emerge as important predictors of HIV-free survival.

METHODOLOGY

We propose to validate the use of a cross-sectional community survey to estimate PMTCT program effectiveness in a predominately rural African setting. The unit of measurement will be at the community level, where we will obtain HIV-free survival estimates using two approaches. Estimates from the community survey will be compared against those of our gold standard community cohort, with statistical correlation and inter-method agreement determined. This study will be implemented within the context of the Better Health Outcomes through Mentoring and Assessment (BHOMA) evaluation, conducted by locally by Zambia AIDS Related Tuberculosis (TB) Project (ZAMBART) and collaborating partners (University of Zambia Biomedical Research Ethics Committee (UNZA BREC) Ref# 004-12-08). The roll-out of BHOMA services occurred in a staggered fashion across 42 of 48 health facilities in Chongwe (n=21), Kafue (n=14), and Luangwa Districts (n=7). The community survey evaluation and the community outreach component of BHOMA target the surrounding catchment area for each health facility. Excluded from this evaluation are hospitals, which typically receive referrals from across the district, and military health posts.

Community survey component

We will work to integrate our PMTCT survey methodology into ongoing BHOMA evaluation activities. In each round, individuals are surveyed using a stratified cluster sampling, where the catchment areas serve as the strata. Within each stratum, geographically defined grid squares are randomly sampled. All households in the selected grid square are visited by a survey team, which comprises at minimum a trained research assistant and a clinician. All individuals in the household are enumerated using a personal digital assistant uploaded with a standard enumeration form. The household location is logged using Global Positioning System (GPS) coordinates, which confirms the position to be within the grid square. Enumerated adults present at the home are asked to provide written informed consent to participate in the survey. Older children and adolescents provide assent; younger children and infants require consent of a parent or guardian. Three questionnaires have been developed and implemented: the household, men's, and women's questionnaires. All have been adapted from the standard Demographic and Health Survey and the Sexual Behavior Survey used in Zambia for over a decade. The household questionnaire is completed by the head of household; the men's and women's questionnaires are administered to all adult men and women, respectively, who are home at the time of the visit. In addition, data are collected on participant weight, height, and abdominal circumference; hypertension screening is provided using a digital sphygmomanometer; and voluntary counseling and testing for HIV is offered using sequential testing algorithms endorsed by the Zambian Ministry of Health. HIV results are available in the field and will be disclosed to participants willing to learn their HIV status. Post-test counseling is provided by certified providers at the household and appropriate referrals made.

In this component, we will implement a PMTCT evaluation module to target women reporting a live birth over the past 24 months within the BHOMA survey.

Although HIV testing is offered to adults as part of the main BHOMA survey, we will also collect dried blood spots (DBS) specimens from both mother and infant and link them using pre-printed bar codes. For a mother who refuses real-time testing, but agrees to collection of this maternal DBS specimen, she will be provided a card with a unique study-generated identification number that can be used pick-up results (with appropriate post-test counseling) at the community's designated health facility. For those who agreed to on-site HIV testing, we will retain the DBS specimens for quality assurance purposes. On a regular basis, randomly selected anonymized specimens will be analyzed using ELISA HIV antibody testing. If a high level of discordancy between the on-site rapid test and the lab-based ELISA HIV test is observed, we will test all specimens to confirm maternal HIV status. As part of the informed consent process, participants will also be asked whether leftover specimens may be used for future use, pending local and international ethical approvals for specified substudies.

If the household reports a delivery within the past 24 months, but the mother has died, we will collect as much relevant antenatal, delivery, and postpartum information as possible from the guardian or caretaker. An abbreviated verbal autopsy instrument will be administered to determine whether the cause of death may have been HIV-related. If the infant is still alive, we will collect a DBS specimen via heelstick for HIV antibody testing and possibly HIV DNA PCR. If the infant has died, this will be documented and included as a study event.

Specimens from HIV-exposed infants < 18 months will be tested for HIV infection using HIV DNA PCR. For those who agree at time of informed consent, we will dispatch trained lay counselors to the household to discuss HIV test results, provide post-test counseling, and make any necessary clinic referrals, including for long-term HIV care and treatment.

Community cohort component

To calculate "gold standard" estimates of 18-month HIV-free survival, we will enroll and follow cohorts of HIV-exposed children (and their HIV-infected mothers) for 18 months. To minimize selection biases that may result from facility-based recruitments, we will enroll within the catchment area surrounding the health facility. In each of these communities, we will identify and train community-based research assistants (CRAs) to recruit participants into our community cohorts. To ensure continuity with the government health system, where possible, these individuals will be preferentially recruited from the Neighborhood Health Committees at each facility. We will use facility- and community-based reporting systems from BHOMA to identify all recent births and, within the first 4 weeks of life, approach mothers at their homes to explain the study. Interested candidates will be asked to show written documentation of their HIV status, preferably from their take-home antenatal record. For those without this documentation, we will obtain consent for HIV screening and provide testing on-site using Ministry of Health-approved algorithms. Those who test HIV-negative will be provided routine post-test counseling and referred to the nearest health facility for routine postpartum care. Women who test HIV-positive and those with documented HIV infection from antenatal care will have the study explained to them and asked to provide written informed consent for themselves and their infants to participate.

At initial enrollment, a questionnaire will be administered, including demographic and socioeconomic characteristics, basic medical history, recent obstetrical history, and detailed questions regarding HIV, including PMTCT service utilization in the last pregnancy. Where possible, we will incorporate questions verbatim from the PMTCT evaluation module of the community survey, to ensure comparability between the two populations. A DBS specimen will be collected from the infant for HIV DNA PCR testing.

Following enrollment, three additional household visits are planned: at 6 weeks, 6 months, 12 months, and 18 months. CRAs will complete a short questionnaire focused on ongoing PMTCT interventions and child health (including morbidity and mortality). If available, we will review the Under-5 Card, a take-home medical record for children less than 5 years of age, to further detail the child's medical course. At 6 weeks, 6 months, and 12 months, DBS specimens will again be collected via heelstick for HIV DNA PCR testing. At 18 months, a rapid antibody test will be performed on site. Test results will be returned to the mother at site of her choosing, either at the home or the health facility, by a trained counselor. Children who test HIV-positive will be referred to the nearest health facility for confirmation of the diagnosis and for long-term care.

Facility survey component

Study staff will complete detailed facility survey questionnaires at all 42 facilities. They will administer a modified version of "A Rapid Health Facility Assessment Tool: to Enhance Quality and Access at the Primary Health Care Level". The instrument comprises four modules: a quality-of-care checklist completed under direct observation of first antenatal visits (Module 1); an exit interview with up to six consecutive pregnant women to measure knowledge and perception about clinical care (Module 2); a checklist of available supplies and infrastructure on site (Module 3); and an interview with the facility manager regarding services provided, staffing levels, and facility descriptors (Module 4). In addition, a time-motion component records the waiting time between registration and patient encounter, duration of the total visit, and duration of post-test counseling.

Prior to implementation, we will field-test the survey instrument in focus groups and refine it as needed. Based on limitations identified from our previous analysis, we expect to increase the number of directly observed patient encounters from six to 15-20 individuals and standardize the type of visits encountered. We may also consider completion of the facility survey over multiple site visits, so that responses from a single clinic visit is not given undue weight. All data will be entered into a Microsoft Access database and seven facility performance scores - again, based on the previous PEARL study - will be calculated based on a priori groupings of characteristics: antenatal care, PMTCT, supplies, staffing levels, patient satisfaction, general infrastructure, and patient understanding of medications. Both individual characteristics and composite scores will be compared against the outcome of HIV-free survival.

ELIGIBILITY:
Eligibility criteria for community cohort:

* We will use facility- and community-based reporting systems from BHOMA to identify all recent births and, within the first 4 weeks of life, approach mothers at their homes to explain the study. Mothers are screened for HIV status, by on-site test and by medical record review (if available)

Eligibility criteria for community survey:

* We will enrollment HIV-infected women who report a delivery of an infant in the past 24 months

Max Age: 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: HIV-infected women and their HIV-exposed infants / children
Sampling Method: Non-Probability Sample
Enrollment: 827 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HIV-free survival among HIV-exposed infants. | 18 months
  Our primary outcome will be HIV-free survival at 18 months among HIV-exposed infants. HIV-free survival has been proposed as a more comprehensive measure of PMTCT program effectiveness than HIV infections alone, since health services may have a broader health impact outside of interrupted transmission. We have chosen the 18-month time point for several reasons. Because the vast majority of HIV-exposed infants will have stopped breastfeeding by this age, this will provide more complete ascertainment of mother-to-child transmission compared to earlier measurements. This time point has also been endorsed by the WHO as one of two priority outcomes for PMTCT impact evaluations. Since both methodologies will sample and recruit participants from within the community, our measures will be population-based (vs. facility-based).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chi, MD, Principal Investigator — UNC at Chapel Hill, Center for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Reseach in Zambia, Lusaka, Zambia